CLINICAL TRIAL: NCT00367978
Title: A Randomized, Multicenter, Study to Determine the Efficacy and Safety of Amlodipine/Benazepril Hydrochloride Versus Enalapril in the Treatment of Hypertension in an African-American Population With Type 2 Diabetes
Brief Title: Effects of Amlodipine/Benazepril in the Hypertensive African-American Population With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCIB002FUS06
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2006-08

CONDITIONS: Hypertension
Keywords: Hypertension, diabetes, African-American, amlodipine/benazepril
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — benazepril

INTERVENTIONS:
Drug: Amlodipine/benazepril

SUMMARY:
This study evaluated the efficacy and safety of amlodipine/benazepril compared with that of enalapril in the treatment of hypertension in African-American patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* African-American
* males and females
* current diagnosis of type 2 diabetes documented by medical history;
* mean sitting diastolic blood pressure of ≥ 90 and ≤ 110 mm Hg;
* HbA1C ≤ 9.5%

Exclusion Criteria:

* having unilateral or bilateral renal artery stenosis;
* having clinically significant cardiac dysrhythmias;
* having a significant history of coronary artery disease within the past 6 months;
* having a history or diagnosis of congestive heart failure (CHF);
* having any clinically relevant cardiac valvular disease

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2001-12; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Time from baseline to the achievement of first treatment success (defined as achieving a blood pressure (BP) <130/80 mm Hg). The proportion and cumulative proportion of patients who achieved first treatment success were also determined.

SECONDARY OUTCOMES:
change from baseline in sitting diastolic BP at Week 24
change from baseline in sitting systolic BP at Week 24
change from baseline in urinary protein excretion at Week 24
change from baseline in HbA1c at Week 24
change from baseline in estimated glomerular filtration rate (EGFR) at Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Corporation, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals Corporation, East Hanover, New Jersey, United States